CLINICAL TRIAL: NCT04249999
Title: A Randomised Controlled Trial of a Novel Web-based Intervention to Promote Physical Activity Participation in People With Cystic Fibrosis
Brief Title: ActivOnline: Physical Activity in Cystic Fibrosis Trial UK
Acronym: ActiOnPACTUK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: University of Exeter (Other)
Collaborators: Cystic Fibrosis Trust (Other); Sport England (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1819/04
Record Dates: First submitted 2019-11-13; First posted 2020-01-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Masking Description: Physical activity intervention. Assignment to intervention or control group cannot be blinded.
  Follow-up assessments will be conducted by blinded assessors.
  UPADTE JUNE 2021: As noted in update above, all participants will perform procedures themselves within their own homes (i.e. physical activity, lung function, questionnaires). Therefore, use of blinded assessors is no longer applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to online physical activity platform (www.activonline.com.au) in addition to usual care.
  Interventions: Behavioral: ActivOnline
- Control (No Intervention): No access to online physical activity platform. Continue with usual care.

INTERVENTIONS:
Behavioral: ActivOnline — Access to online physical activity platform (www.activonline.com.au)
  Arms: Intervention

SUMMARY:
Increased level of physical activity (PA) are of benefit in the management of cystic fibrosis (CF). This randomised control tial will assess whether three-months use of an online platform can help increase PA levels in people with CF (compared to a control group continuing routine treatment).

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic condition that predominantly affects the lungs through an accumulation of thick mucus. As there is no cure for CF, it is a disease that is managed through intensive medication, nutrition, physiotherapy, exercise and physical activity (PA).

Increased levels of PA are of benefit to people with CF, and therefore interventions that promote PA are warranted, particularly in adolescence, whereby PA levels decrease. Telehealth interventions are of particular interest in CF, whereby strict cross-infection guidelines prevent patients meeting in person, and allowing patients to overcome geographical barriers at the same time.

Previous research has shown engagement with an online platform (www.activonline.com.au), specifically designed to monitor PA in CF, is feasible and acceptable to people with CF. Therefore, a full randomised control trial is warranted to assess the efficacy of this intervention in changing PA.

UPDATE JUNE 2021: Due to ongoing restrictions placed upon research by the global COVID-19 pandemic, modifications to the protocol are necessary.

Recruitment and consenting will now take place online, and testing procedures will be completed by participants in their own homes. The nature, and length of, intervention remains unchanged.

Changes to protocol approved by ethics board on May 4th 2021.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* Aged 12-35 years (inclusive)
* Able to provide informed consent/assent
* Able to access the internet via computer or mobile device

Exclusion Criteria:

* Presence of severe co-morbidity limiting mobilisation or physical activity participation (e.g. orthopaedic, cardiac or neurological condition)
* Previous lung transplantation
* Pregnancy
* Unable to provide informed consent/assent

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity, objectively measures using ActiGrpah GT9X Link accelerometer. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Time spent in sedentary, light, moderate and vigorous physical activity domains will be assessed over a one week period. Accelerometer to be worn on non-dominant wrist.
Change in physical activity, subjectively measured using the Habitual Activity Estimation Scale. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Questionnaire determines time spent being inactive, somewhat inactive, somewhat active and very active, each reported as a percentage of the day.

SECONDARY OUTCOMES:
Change in forced expiratory volume in one second (FEV1), measured in absolute units (L) | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Assessment of lung function
Change in forced vital capacity (FVC), measured in absolute units (L) | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Assessment of lung function
Change in forced expiratory volume in one second (FEV1), measured as a percent of predicted, as per GLI2012 equations. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Assessment of lung function
Change in forced vital capacity (FVC), measured as a percent of predicted, as per GLI2012 equations. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Assessment of lung function
Change in exercise attitudes, measured using the Behavioural Regulation in Exercise Questionnaire. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Assessment of reasons underlying people's decision to engage, or not engage, in exercise. Scores range from -24 to +20, where a higher score indicates greater exercise autonomy (better outcome).
Change in quality of life, measured using age-specific Cystic Fibrosis Questionnaire (Revised). | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Subjective assessment of health related quality of life, scored from 0 to 100 where a higher score indicates higher quality of life (better outcome).
Change in anxiety, measured using Hospital Anxiety and Depression Scale. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Subjective report of anxiety, scored from 0 to 21, where a higher score indicates higher anxiety (worse outcome).
Change in depression, measured using Hospital Anxiety and Depression Scale. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Subjective report of depression, scored from 0 to 21, where a higher score indicates higher depression (worse outcome).
Change in depression, measured using Center for Epidemiological Studies-Depression Scale. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Subjective reports of anxiety and depression, scored from 0 to 60 where a higher score indicates greater depressive symptoms (worse outcome).
Change in sleep quality, measured using Pittsburgh Sleep Quality Index (PSQI). | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks).
  Subjective report of sleep quality, scored from 0 to 21 where a higher score indicates worse sleep quality (worse outcome).

OTHER OUTCOMES:
Qualitative assessment of barriers and facilitators to physical activity | 3-months post-intervention (+24 weeks)
  Semi-structured, 10-item interview for participants in both intervention and control group
Qualitative assessment of Activ Online programme | 3-months post-intervention (+24 weeks)
  Semi-structured interview question for participants assigned to intervention group
Usage of Activ Online programme | Post-intervention (+12 weeks)
  Frequency of access and logging of physical activity data
Changes in physical activity, measured by Sport England Short Active Lives Survey. | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks)
  Subjective assessment of physical activity
Changes in physical activity, measured by Sport England Engagement in Sport Questions | Baseline, post-intervention (+12 weeks), 3-months post-intervention (+24 weeks)
  Subjective assessment of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Williams, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox NS, Alison JA, Button BM, Wilson JW, Holland AE. Feasibility and acceptability of an internet-based program to promote physical activity in adults with cystic fibrosis. Respir Care. 2015 Mar;60(3):422-9. doi: 10.4187/respcare.03165. Epub 2014 Nov 25. PMID 25425703
- [Background] Cox NS, Eldridge B, Rawlings S, Dreger J, Corda J, Hauser J, Button BM, Bishop J, Nichols A, Middleton A, Ward N, Dwyer T, Tomlinson OW, Denford S, Barker AR, Williams CA, Kingsley M, O'Halloran P, Holland AE; Youth Activity Unlimited - A Strategic Research Centre of the UK Cystic Fibrosis Trust. A web-based intervention to promote physical activity in adolescents and young adults with cystic fibrosis: protocol for a randomized controlled trial. BMC Pulm Med. 2019 Dec 19;19(1):253. doi: 10.1186/s12890-019-0942-3. PMID 31856791
- [Result] Tomlinson OW, Barker AR, Denford S, Williams CA. Adapting, restarting, and terminating a randomised control trial for people with cystic fibrosis: Reflections on the impact of the COVID-19 pandemic upon research in a clinical population. Contemp Clin Trials Commun. 2024 Mar 27;39:101294. doi: 10.1016/j.conctc.2024.101294. eCollection 2024 Jun. PMID 38577655